CLINICAL TRIAL: NCT00362700
Title: An Open-Label, Phase II Study to Evaluate Safety, Tolerability, Antiviral Activity and Biochemical and Immunological Responses of Retreated Clevudine in Chronic Hepatitis B Patients Who Received Clevudine in L-FMAU-201
Brief Title: Safety and Efficacy Study of Retreated Clevudine in Chronic HBV Patients Who Received Clevudine in L-FMAU-201
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L-FMAU-204
Record Dates: First submitted 2006-08-08; First posted 2006-08-10 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2006-06

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — clevudine

INTERVENTIONS:
Drug: Clevudine

SUMMARY:
The purpose of this study is to determine the safety and antiviral activity of Clevudine, when retreated to patients previously treated with Clevudine

ELIGIBILITY:
Inclusion Criteria:

1. Patients who received clevudine in L-FMAU-201 clinical trial (phase IIb)
2. Female of childbearing potential must have a negative serum ( b-HCG) pregnancy test within 14 days of starting therapy.
3. Patient is able to give written informed consent prior to study start and to comply with the study requirements.
4. Patients who met the following criteria after completion of the Week 48 visit were to have additional follow-up visits at Weeks 54 and 60: 1) had received no additional therapy since completion of 24-week treatment of clevudine and 2)experienced a > 1 log10 decrease from baseline in HBV DNA at Week 48

Exclusion Criteria:

1. HBV DNA negative (< 4,700 copies/mL) consistently at the last 2 visit (at least 2 consecutive visits, at one month interval)
2. Patient is currently receiving antiviral immunomodulatory or corticosteroid therapy.
3. Patients previously treated with lamivudine, lobucavir, adefovir or any other investigational nucleoside for HBV infection after cessation of treatment in L-FMAU-201 study.
4. Patient has a history of ascites, variceal hemorrhage or hepatic encephalopathy.
5. Patient is coinfected with HCV, HDV or HIV.
6. Patient with clinical evidence of cirrhosis or hepatocellular carcinoma (®-Fetoprotein) Evaluation will be based on alpha-fetoprotein primarily. If alpha-fetoprotein level is suggestive of cirrhosis or hepatocellular carcinoma, confirmation will be made with sonography etc.
7. Patient is pregnant or breast-feeding.
8. Patient is unwilling to use an "effective" method of contraception during the study and for up to 3 months after the use of study drug ceases. For males, condoms should be used. Females must be surgically sterile (via hysterectomy or bilateral tubal ligation), post-menopausal or using at least a medically acceptable barrier method of contraception (i.e., IUD, barrier methods with spermicide or abstinence)
9. Patient has a clinically relevant history of abuse of alcohol or drugs.
10. Patient has a significant gastrointestinal, renal, hepatic (decompensated), bronchopulmonary, neurological, cardiovascular, oncologic or allergic disease.
11. Patient has creatinine clearance less than 60mL/min as estimated by the following formula:

(140-age in years) (body weight [kg])/(72) (serum creatinine [mg/dL]) [Note: multiply estimates by 0.85 for women]

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33
Dates: Start 2003-07; Study Completion 2005-10

PRIMARY OUTCOMES:
Antiviral activity- Change from baseline in HBV DNA (log10)
Safety- Laboratory tests, Adverse Events, Vital Signs, ECG

SECONDARY OUTCOMES:
Antiviral activity- Proportion of patients with HBV DNA below the assay Limit of Detection(<4,700 copies/mL by Digene Hybrid Capture II)
Biochemical improvement (ALT normalization)
Serology: Proportion of patients with HBeAg loss,Seroconversion rate (HBeAg loss and anti-HBe gain)

CONTACTS AND LOCATIONS:
Overall Officials: Hyo Suk Lee, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (7):
- South Korea (7):
  - Korea University Guro Hospital, Seoul, Guro-gu
  - Seoul National University Hospital, Seoul, Jongno-Gu
  - Yongdong Severance Hospital, Dogok-dong, Kangnam-gu, Seoul
  - Samsung Medical Center, Ilwon-dong, Songpa-gu, Seoul
  - Ehwa Womans University Mokdong Hospital, Mok-dong, Yangcheon-gu, Seoul
  - Seoul Asan Medical Center, Pungnap-dong, Kangnam-gu, Seoul
  - Asan Medical Center, P’ungnabi-dong, Songpa-Gu, Seoul